CLINICAL TRIAL: NCT00593346
Title: Evaluation of Accelerated Partial Breast Brachytherapy as the Sole Method of Radiation Therapy for Stage 0, 1 and II Lymph Node Negative Breast Carcinoma
Brief Title: Evaluation of Accelerated Partial Breast Brachytherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-1205 / 201011816
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accelerated partial breast brachytherapy (Experimental): Each patient will receive accelerated partial breast brachytherapy with multiple plane implant.
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — brachytherapy (radioactive implants)

SUMMARY:
Over the past two decades, breast conserving therapy (BCT) has become a major treatment modality for Stage I and II breast carcinoma. The major advantages of breast conserving therapy are superior cosmetic outcome and the reduced emotional and psychological trauma afforded by this procedure compared with conventional mastectomy. The principal disadvantage of BCT is its more complex and prolonged treatment regimen requiring approximately 6 weeks of external beam radiation therapy that poses problems for some patients such as the working woman, elderly patients, and those who live at a significant distance from a treatment center. These factors, along with the patient's geographic location, result in a smaller fraction of the patients who currently meet eligibility criteria for BCT actually receiving it, despite its cosmetic and probable psychological advantages. The logistical problems of BCT are primarily related to the protracted course of external beam radiation therapy to the whole breast. While some investigators reported what they believe to be acceptable local control rates in carefully selected patients treated by wide local excision without radiation therapy, the criteria for patient selection are controversial and poorly defined and probably restrict the access of many patients to breast conserving therapy.

If previous observations are valid and breast irradiation following tylectomy exerts its maximal effect in eradicating occult disease remaining in the immediate vicinity of the tylectomy site, can radiation therapy be directed only to the tissue surrounding the excision cavity of the breast, using brachytherapy alone? If so, the entire course of radiation therapy could be delivered over a 4 to 7 day period immediately following tylectomy and/or axillary dissection, thus markedly reducing treatment time. Brachytherapy also inherently provides a higher central dose to the volume most at risk for recurrence. Cosmetic outcome after the use of a brachytherapy boost after external whole breast radiotherapy is comparable or slightly inferior to electron beam boost radiation therapy

DETAILED DESCRIPTION:
This study will evaluate the local control, cosmetic results, quality of life, and complication rates of brachytherapy when used as the sole method of radiation therapy for patients with stage 0,I, and II carcinoma of the breast treated with tylectomy, with histologically assessed negative surgical margins, N0 axillary nodes.

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage 0, I, or II (TisN0, T1N0, T2N0 = 3 cm) histologically confirmed carcinoma of the breast, treated with tylectomy. Axillary sampling is required only for cases of invasive cancers. Tumor size is determined by the pathologist. Clinical size may be used if the pathologic size is indeterminate.
* Signed study-specific informed consent for participation in the study.
* Negative, or close but negative, inked histologic margins of tylectomy or reexcision specimen to be confirmed prior to placing the brachytherapy catheters. Margins generally are positive if there is invasive or noninvasive tumor at the inked resection margin, close but negative if the tumor is within 2 mm of the inked margin and negative if the tumor is at least 2 mm away from the inked edge.
* Negative post-tylectomy or post-reexcision mammography if cancer presented with malignancy-associated microcalcifications; no remaining suspicious microcalcifications in the breast before brachytherapy.
* For patients with invasive cancer, no positive axillary lymph nodes with at least 6 axillary lymph nodes sampled or a negative sentinel node.
* Invasive ductal, lobular, medullary, papillary, colloid (mucinous),or tubular histologies. Noninvasive ductal carcinoma in situ.
* Chemotherapy or hormonal therapy planned for = 2 weeks after removal of brachytherapy catheters is permitted. Hormonal therapy is allowed during brachytherapy at treating radiation oncologist's decision.
* Negative pregnancy test for premenopausal patients with an intact uterus

Exclusion Criteria:

* Patients with distant metastases.
* Patients with in-situ lobular carcinoma or nonepithelial breast malignancies such as sarcoma or lymphoma.
* Patients with proven multicentric carcinoma (tumors in different quadrants of the breast, or tumors separated by at least 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy.
* Patients who are pregnant or lactating.
* Patients with histologically confirmed positive axillary nodes in the ipsilateral axilla. Palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
* Prior non-hormonal therapy for the present breast cancer, including radiation therapy or chemotherapy.
* Patients with systemic lupus erythematosis, scleroderma, or dermatomyositis with a CPK level above normal or with an active skin rash.
* Patients with coexisting medical conditions in whom life expectancy is < 2 years.
* Patients with psychiatric or addictive disorders that would preclude obtaining informed consent or completing the full series of high dose rate brachytherapy treatments on an outpatient basis.
* Patients with Paget's disease of the nipple.
* Patients with skin involvement, regardless of tumor size.
* Patients with a breast unsatisfactory for brachytherapy. For example, if there is little breast tissue remaining between the skin and pectoralis muscle after surgery, placement of catheters is technically problematic.
* Patients with tylectomies so extensive that the cosmetic result is fair or poor prior to brachytherapy.
* Surgical margins which cannot be microscopically assessed or are positive at pathological evaluation.
* Any previously treated contralateral breast carcinoma or synchronous bilateral breast carcinoma.
* Other malignancy, except non-melanoma skin cancer, ≤ 5 years prior to participation in this study; the disease free interval from any prior carcinoma must be continuous.
* Time between final definitive breast procedure to radioactive source loading of the brachytherapy catheters is greater than 8 weeks.
* Patients with diffuse (> 1 quadrant or >5 cm in diameter) suspicious microcalcifications.
* Patients with suspicious microcalcifications remaining on the post-tylectomy mammogram

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2004-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on March 12, 2004 and closed to participant enrollment on 12/22/2008.
Groups:
- Accelerated Partial Breast Bracytherapy: Each patient will receive accelerated partial breast brachytherapy with multiple plane implant.
  Patients will receive 3400 cGy delivered in 10 twice-daily fractions. Treatment is to be given over 5-7 days with a minimum of 6 hours separation between fractions.
Period: Overall Study
Arm/Group | Accelerated Partial Breast Bracytherapy
Started | 151
Completed | 151
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Accelerated Partial Breast Brachytherapy: Each patient will receive accelerated partial breast brachytherapy with multiple plane implant.
  Patients will receive 3400 cGy delivered in 10 twice-daily fractions. Treatment is to be given over 5-7 days with a minimum of 6 hours separation between fractions.
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
Age, Continuous [Mean (Full Range); unit: years] | 60 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 151
Race [Number; unit: participants]
  Caucasian | 128
  African-American | 23
Residence at diagnosis [Number; unit: participants]
  Urban area | 111
  Urban cluster | 25
  Rural | 15
Tumor location [Number; unit: participants]
  Upper outer quadrant | 54
  Upper inner quadrant | 46
  Lower outer quadrant | 30
  Lower inner quadrant | 21
Pathologic tumor stage [Number; unit: participants] — Tis: Carcinoma in situ. T1mic: Microinvasive ductal carcinoma T1a: Tumor >1 mm but ≤5 mm in greatest dimension. T1b: Tumor >5 mm but ≤10 mm in greatest dimension. T1c: Tumor >10 mm but ≤20 mm in greatest dimension. T2: Tumor >20 mm but ≤50 mm in greatest dimension.
  participants
    Tis | 28
    T1mic | 1
    T1a | 19
    T1b | 52
    T1c | 38
    T2 | 13
Sentinel lymph node biopsy [Number; unit: participants] — Only for patients with invasive cancer
  participants
    Yes | 122
    No | 1

OUTCOME MEASURES:

1. Primary Outcome: Local Control Using Ipsilateral Breast Tumor Recurrence Rates
Time Frame: 2 years after treatment completion
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
percentage of participants | .7

2. Secondary Outcome: Quality of Life Completion
Description: -QOL was assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and EORTC breast cancer module QLQ-BR23 questionnaires. QLQ-C30 is composed of 30 questions. QLQ-BR23 consists of 23 questions.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
percentage of participants
  6-8 weeks | 99
  3-4 months | 95
  6-8 months | 91
  1 year | 88
  2 years | 74

3. Secondary Outcome: Excellent-good Cosmetic Outcomes - Patient Reported
Description: * Both the participants and the treating radiation oncologist qualitatively rated cosmesis as excellent, good, fair, or poor over time and ascribed a cause for changes in cosmesis.
  * The global cosmetic result were scored on a 4-point scare where 0=excellent result (no difference), 1=good (small difference), 2=fair result (moderate difference) and 3=poor result (large difference).
Time Frame: 3 years after completion of therapy
Population: 82 participants had cosmetic outcome data through 3 years of follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 82
percentage of participants
  Pre-treatment | 92
  3-4 months after treatment | 91
  2 years | 87
  3 years | 92

4. Secondary Outcome: Excellent-good Cosmetic Outcomes - Physician Reported
Description: * Both the participants and the treating radiation oncologist qualitatively rated cosmesis as excellent, good, fair, or poor over time and ascribed a cause for changes in cosmesis. Cosmetic outcome was evaluated quantitatively by percentage of breast retraction assessment (pBRA).
  * The global cosmetic result were scored on a 4-point scale where 0=excellent result (no difference), 1=good (small difference), 2=fair result (moderate difference) and 3=poor result (large difference).
Time Frame: 3 years after completion of therapy
Population: 82 participants had cosmetic outcome data through 3 years of follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 82
percentage of participants
  Pre-treatment | 97
  3-4 months after treatment | 97
  2 years | 94
  3 years | 94

5. Secondary Outcome: Impressions of the Cause of Cosmesis Changes Over Time - Patient Reported
Description: -Patients filled out a form "Patient Evaluation of the Treated Breast". On this form the patients were asked to compare the memory of what their breast looked like after surgery but before radiation and to compare that memory to the appearance of the breast after radiation. The patients were then asked if their breast changes were due to:
  * caused mostly by radiation
  * caused by both the radiation and surgery, but mostly by the radiation
  * caused by both the radiation and surgery, but mostly by the surgery
  * caused mostly by the surgery
  * can't judge which treatment caused the change
  * there are no changes
Time Frame: 3 years
Population: 82 participants had cosmetic outcome data through 3 years of follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 82
percentage of participants
  Radiation | 16.5
  Surgery | 57
  Unsure | 19
  No cosmetic changes | 7.5

6. Secondary Outcome: Cosmesis Outcome as Measured by Percentage of Breast Retraction Assessment (pBRA)
Description: -Cosmetic outcome was evaluated quantitatively by percentage of breast retraction assessment (pBRA)
Time Frame: Pre-treatment and 3 years
Population: 82 participants had cosmetic outcome data through 3 years of follow-up.
Measure: Mean (95% Confidence Interval); unit: percentage of breast retraction
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 82
percentage of breast retraction
  Pre-treatment | 7.35 [6.49 to 8.21]
  3 years | 7.64 [6.68 to 8.6]

7. Primary Outcome: Local Control as Measured by Ipsilateral Breast Tumor Recurrence Rates
Time Frame: 5 years after treatment completion
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
percentage of participants | 3.4

8. Primary Outcome: Local Control Using Disease-free Survival Rates
Time Frame: 2 years after treatment completion
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
percentage of participants | 99.3

9. Primary Outcome: Local Control Using Disease-free Survival Rates
Time Frame: 5 years after treatment completion
Measure: Number; unit: percentage of participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
percentage of participants | 94.4

10. Secondary Outcome: Presence or Absence of Complications
Description: As defined by number of participants who experienced breast infection and symptomatic fat necrosis.
Time Frame: 5 years after treatment completion
Measure: Number; unit: participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
participants
  Breast infection | 6
  Fat necrosis (symptomatic) | 19

11. Secondary Outcome: Occurrence of Mastectomy After Completion of Initial Breast-conserving Treatment
Time Frame: 5 years after treatment completion
Measure: Number; unit: participants
Arm/Group | Accelerated Partial Breast Bracytherapy
Number analyzed (Participants) | 151
participants | 4

12. Secondary Outcome: Frequency of Grade 3-4 Toxicities
Description: RTOG acute and late toxicity grading system and via a visual analog scale for pain assessment.
Time Frame: Up to 1 year from completion of therapy
Measure: Number; unit: participants
Arm/Group | Accelerated Partial Breast Brachytherapy
Number analyzed (Participants) | 151
participants
  Acute skin - Grade 3/4 | 1
  Acute breast infection - Grade 3/4 | 2
  Acute subcutaneous - Grade 3/4 | 0
  Late skin - Grade 3/4 | 0
  Late subcutaneous | 0
  Late heart - Grade 3/4 | 0
  Late pulmonary - Grade 3/4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment through 1 year after completion of treatment.
Arm/Group | Accelerated Partial Breast Bracytherapy
Serious Adverse Events (participants affected / at risk) | 0/151
Other Adverse Events (participants affected / at risk) | 151/151
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accelerated Partial Breast Bracytherapy (N=151)
Acute skin (Skin and subcutaneous tissue disorders) | 58
Acute breast infection (Infections and infestations) | 6
Acute subcutaneous (Skin and subcutaneous tissue disorders) | 13
Late skin (Skin and subcutaneous tissue disorders) | 36
Late subcutaneous (Skin and subcutaneous tissue disorders) | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes